CLINICAL TRIAL: NCT00957567
Title: A Comparison Study of Breast Tomosynthesis Images Reconstructed at 1 Millimeter and 5 Millimeter Slice Thicknesses
Brief Title: Comparison Study of Breast Tomosynthesis Slice Thicknesses
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Principal Investigator, Mary Newell, MD, Associate Professor, Emory University
Other Study IDs: IRB00008667
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Early diagnosis is one of the most important factors in the survival of patients diagnosed with breast cancer. To aid in the early detection of breast cancer, a new technology, called tomosynthesis imaging is being developed. The idea behind tomosynthesis imaging is to "look" at the breast from different points of view by obtaining x-ray flat images from different angles while the breast does not move, and then mathematically combine these flat images into a three-dimensional image. The benefit of these three dimensional images is that the radiologist can look at the different tissues of the breast in their real positions, as opposed to all the tissues being "flattened" into a flat image, like that of a normal mammogram. Since tomosynthesis images of the breast show the tissues in their real position, the radiologist should be able to more easily find a tumor and also be able to reduce the number of time he or she thinks there is a tumor present when in reality there is not one there.

Before this new technology can be used in the clinic routinely, it is necessary to perform a large number of studies to find the optimal way to use it. In this study, the investigators are aiming to find how thick the slices or layers representing the breast should be in the image when shown to the radiologist. The difference between these two thicknesses in how useful the images are to the radiologist could be important. The investigators are trying to determine if slicing the image of the breast into thicker slices will make the job of the radiologist easier or not when deciding to recommend or not a biopsy (laboratory analysis) of what the previous mammogram found. To find the answer to this question, the investigators will image patients with their tomosynthesis machine and look at the tomosynthesis images with the thin and thick slices. The radiologists that read each image will decide if they would have recommended the patient to get a biopsy based only in each of these images. The recommendations based on the images with thin slices and the recommendations based on the images with thick slices will be compared with what was actually recommended using the standard clinical tests. The investigators hope to find that the thicker slices help more than the thinner slices when trying to decide if biopsy is needed or not.

DETAILED DESCRIPTION:
Early diagnosis is one of the most important factors in the survival of patients diagnosed with breast cancer. To aid in the early detection of breast cancer, a new technology, called tomosynthesis imaging is being developed. The idea behind tomosynthesis imaging is to "look" at the breast from different points of view by obtaining x-ray flat images from different angles while the breast does not move, and then mathematically combine these flat images into a three-dimensional image. The benefit of these three dimensional images is that the radiologist can look at the different tissues of the breast in their real positions, as opposed to all the tissues being "flattened" into a flat image, like that of a normal mammogram. The flat images in mammograms bring about the possibility that normal healthy tissue sometimes covers up malignant tumors, making them harder, and sometimes impossible, for the physician to see. In addition, this "flattening" sometimes generates what appears to be suspicious tissue, but is in reality a superposition of normal healthy tissue. This effect results in performing an increased number of biopsies that end up being negative for breast cancer. Since tomosynthesis images of the breast show the tissues in their real position, these effects can be avoided. It has already been shown by various research labs, including ours, that this kind of imaging does in fact result in better visualization of lesions compared to conventional two-dimensional imaging, even without performing tomosynthesis under ideal conditions.

For tomosynthesis to reach its full potential, it is necessary to perform a large number of studies to find the optimal way to acquire the tomosynthesis images and the optimal way to mathematically combine these images to get the three dimensional image. In this study, we are aiming to find if the resulting three dimensional image should be divided into slices or layers each representing 1 millimeter (less than one 16th of an inch) of the breast or 5 millimeters (one 5th of an inch) of the breast. The difference between these two thicknesses in how useful the images are to the radiologist could be important. Up to now, tomosynthesis imaging has been performed with 1 millimeter slices, but there has been no scientific study to prove that this is the best slice thickness. We will try to determine if slicing the image of the breast into thicker slices will make the job of the radiologist easier or not when deciding to recommend or not a biopsy (laboratory analysis) of what the previous mammogram found. To find the answer to this question, we will image patients with our tomosynthesis machine and look at the tomosynthesis images with the thin and thick slices. The radiologists that read each image will decide if they would have recommended the patient to get a biopsy based only in each of these images. The recommendations based on the images with thin slices and the recommendations based on the images with thick slices will be compared with what was actually recommended using the standard clinical tests. We hope to show that the images with the thick slices will do as well if not better than those with the thin slices. Even if the thick slices only do as well as the thin slices, this will show that creating images with thicker slices is better, since these images can be read faster by the radiologist.

ELIGIBILITY:
3.1 Eligibility Criteria All subjects will be women at least 35 years of age that have been found, after diagnostic workup, to have focal distributions of microcalcifications (BI-RADS 3, 4 or 5), focal soft tissue lesions (BI-RADS 3, 4 or 5), or no findings (BI-RADS 1).

3.2 Ineligibility Criteria

* Subject does not meet any of the inclusion criteria
* Women with suspected or confirmed pregnancy
* Women who have had bilateral mastectomy
* Women with large breasts that cannot be accommodated within the field of view of the tomosynthesis system
* Women who are very frail and unable to cooperate
* Women who are under 35 years of age
* Women who cannot give informed consent
* Male subjects
* Women with implants
* Subject has had breast augmentation, except for unilateral augmentation done for prior mastectomy

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for this study is women who are recalled for an abnormal finding on a screening mammogram.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Equivalence in diagnostic accuracy | After biopsy or follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mary Newell, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Breast Imaging Center, Atlanta, Georgia, United States